CLINICAL TRIAL: NCT07098104
Title: Identifying Optimal Responders: A Benefit Population Atlas of Neoadjuvant Immunochemotherapy Versus Chemotherapy for Locally Advanced Gastric Cancer
Brief Title: A Benefit Population Atlas of nICT Versus nCT for LAGC
Status: Completed | Type: Observational
Sponsor: Cheng Chen (Other)
Responsible Party: Sponsor-Investigator, Cheng Chen, Associate Chief Physician, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Other Study IDs: KY-2025-066
Record Dates: First submitted 2025-07-27; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immunotherapy; sintilimab; tislelizumab; Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant chemotherapy: The nCT group included two subgroups: nCT2 (SOX/XELOX) and nCT3 (FLOT: docetaxel 50mg/m² + oxaliplatin 85mg/m² + leucovorin 200mg/m² d1 + fluorouracil 2600mg/m² 48h CIV q2w; or DCF: docetaxel 75mg/m² + cisplatin 75mg/m² d1 + fluorouracil 750mg/m² d1-5 q3w).
  Interventions: Drug: Immunotherapy
- neoadjuvant immunochemotherapy: The nICT group received PD-1 inhibitors (sintilimab 200mg, tislelizumab 200mg, or nivolumab 240mg, all iv q3w) combined with two-drug chemotherapy (SOX: oxaliplatin 130mg/m² d1 + S-1 40-60mg bid d1-14; or XELOX: oxaliplatin 130mg/m² d1 + capecitabine 1000mg/m² bid d1-14, both q3w).
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — The nICT group received PD-1 inhibitors (sintilimab 200mg, tislelizumab 200mg, or nivolumab 240mg, all iv q3w) combined with two-drug chemotherapy (SOX: oxaliplatin 130mg/m² d1 + S-1 40-60mg bid d1-14; or XELOX: oxaliplatin 130mg/m² d1 + capecitabine 1000mg/m² bid d1-14, both q3w). The nCT group included two subgroups: nCT2 (SOX/XELOX) and nCT3 (FLOT: docetaxel 50mg/m² + oxaliplatin 85mg/m² + leucovorin 200mg/m² d1 + fluorouracil 2600mg/m² 48h CIV q2w; or DCF: docetaxel 75mg/m² + cisplatin 75mg/m² d1 + fluorouracil 750mg/m² d1-5 q3w).
  Other Names: sintilimab; tislelizumab; nivolumab

SUMMARY:
The purpose of this observational study is to evaluate the impact of different neoadjuvant therapies on patients with locally advanced gastric cancer. The primary question it aims to address is: Which patient populations benefit most from neoadjuvant immunochemotherapy versus neoadjuvant chemotherapy in locally advanced gastric cancer?

DETAILED DESCRIPTION:
This study aims to: 1. Compare pCR rates and TRG between neoadjuvant chemotherapy (two-drug vs. three-drug) and neoadjuvant immunochemotherapy; 2. Explore efficacy differences across subgroups; 3. Provide evidence-based guidance for individualized neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients had pathologically confirmed adenocarcinoma, imaging-confirmed resectable LAGC (cT2-4aN0-3M0, AJCC 8th), no distant metastases, and completed protocol-specified neoadjuvant therapy (nICT: PD-1/PD-L1 inhibitors plus two-drug chemotherapy; nCT: two-drug [SOX/XELOX] or three-drug [FLOT/DCF] chemotherapy) with ECOG 0-1.

Exclusion Criteria:

Exclusion criteria included incomplete neoadjuvant therapy, non-radical surgery, other malignancies, active autoimmune diseases/immunosuppressant use, missing key data, or inadequate follow-up (<3 months without documented events).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study screened 10,334 patients diagnosed with gastric/gastroesophageal junction tumors at a tertiary-grade A cancer hospital from November 2019 to December 2023 , identifying 777 who received neoadjuvant therapy, with 291 meeting inclusion criteria for final analysis. The cohort comprised resectable gastric adenocarcinoma patients undergoing neoadjuvant immunochemotherapy (nICT, n=98) or chemotherapy (nCT, n=193) followed by radical surgery (Figure S1), with follow-up through November 2024.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
PCR | 2019.11-2023.12
  Pathological complete response
TRG | 2019.11-2023.12
  tumor regression grade

SECONDARY OUTCOMES:
OS | 2019.11-2023.12
  overall survival
EFS | 2019.11-2023.12
  event-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided